CLINICAL TRIAL: NCT02835846
Title: Investigation of the Effect of the Female Urinary Microbiome on Incontinence
Acronym: FUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Kimberly-Clark Corporation (Industry)
Responsible Party: Principal Investigator, Alan J. Wolfe, Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 207777
Record Dates: First submitted 2016-07-10; First posted 2016-07-18 (Estimated); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2020-11

CONDITIONS: Overactive Bladder; Incontinence; Nocturia
Keywords: Overactive Bladder Syndrome; Female Urinary Microbiome; Urinary Urgency; Estrogen; Nocturia; Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Estrogen Arm (Experimental): The intervention for this study is an estrogen cream (i.e., Premarin Cream®). Women in this study will receive this estrogen cream and apply it to their vagina twice weekly for 12 weeks
  Interventions: Drug: Estrogen Cream

INTERVENTIONS:
Drug: Estrogen Cream — Participants are provided a vaginal estrogen cream (i.e., Premarin Cream® 0.625 mg conjugated estrogen/gram) and instructed to use 0.5 grams with an applicator twice weekly for 12 weeks.
  Other Names: Premarin Cream®

SUMMARY:
This purpose of this study is to understand the types of bacteria that are in the bladder and vagina in patients with overactive bladder (OAB) symptoms and understand if the types of bacteria change when with the use of estrogen in the vagina. The investigators are also trying to understand how estrogen influences the body's ability to make substances called peptides that can kill bacteria.

DETAILED DESCRIPTION:
Overactive bladder (OAB) syndrome is characterized by the symptom complex of urinary urgency, usually with associated frequency and nocturia, with or without urgency urinary incontinence in the absence of infection or other pathology. OAB affects approximately 31% of women over the age of 65. Vaginal estrogen, a well-documented treatment for OAB in hypoestrogenic women, has been shown to improve symptoms of frequency, urgency and urgency urinary incontinence (UUI). Several theories have been proposed to explain the mechanism underlying estrogen's effect on lower urinary tract symptoms (LUTS). The investigators propose that estrogen treatment influences bacterial communities (microbiomes) in the vagina and bladder and alters urothelial and vaginal (AMPs) thereby improving OAB symptoms in hypoestrogenic women.

Long-standing medical dogma has been replaced by clear evidence that a female urinary microbiome (FUM) exists. The investigators recently reported that the FUM in women without OAB is less diverse than the FUM of women with OAB. The investigators soon will report that FUM status stratifies women with OAB into treatment response groups and women with less diverse FUMs are more likely to respond to anti-cholinergic OAB therapy (Thomas-White et al., in preparation). This suggests that the FUM is a factor in lower urinary tract symptoms (LUTS) and that FUM diversity contributes to LUTS and treatment response, like the vaginal microbiome and its contribution to vaginal symptoms.

In hypoestrogenic women, the vaginal microbiome shifts from low diversity communities, commonly dominated by Lactobacillus, to more diverse communities dominated by anaerobes; this change can be reversed with estrogen treatment. Since the FUM of women with OAB includes bacteria similar to those of the vaginal microbiome (e.g. Lactobacillus, Gardnerella, and diverse anaerobes), the investigators reason the FUM would respond similarly to estrogen and become less diverse. Although transvaginal medications likely alter nearby bacterial niches (e.g. the bladder), no study has reported the urinary microbiomic response to vaginal estrogen.

While almost nothing is known about urinary/vaginal microbiome interplay, even less is known about immune response modulation in the bladder and vagina. However, estrogen reduces the subsequent urinary tract infection (UTI) rate in hypoestrogenic women affected by recurrent UTI, and estrogen induces urothelial antimicrobial peptide (AMP) expression. Since AMPs exhibit microbicidal activity, stimulate inflammation, and facilitate epithelial barrier homeostasis, estrogen may work through AMPs as mediators to optimize microbial equilibrium.

The investigators hypothesize that, following estrogen treatment of hypoestrogenic women with OAB, symptom improvement will be associated with 1) reduced FUM diversity, 2) alteration of other FUM characteristics and 3) increased AMP levels. The investigators propose two specific aims:

Aim 1: To compare pelvic floor microbiome (PFM) diversity and AMP levels before and after estrogen treatment in hypoestrogenic women with OAB symptoms.

Aim 2: Determine if FUM characteristics correlate with OAB symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women who present with symptoms of OAB, defined as a condition characterized by urgency, with or without urgency incontinence, usually with frequency and nocturia in the absence of obvious pathology or infection [9], with atrophic vaginitis.
* Postmenopausal by history (i.e., defined as twelve months or greater since last menstrual period), surgical menopause with removal of bilateral ovaries, or age over 55 with a previous hysterectomy (without removal of bilateral ovaries).
* English language skills sufficient to complete questionnaires
* Clinical indication for vaginal estrogen use (i.e., hypoestrogenic findings on physical examination)
* Patients not currently receiving vaginal estrogen therapy

Exclusion Criteria:

* Patients currently on systemic hormone replacement therapy (HRT) or who have been on HRT within the past three months
* Patients with current diagnosis or history of estrogen dependent malignancies (e.g., breast or endometrial malignancies)
* Contraindication or allergy to estrogen therapy
* Insufficient English language skills to complete study questionnaires
* Women with active, standard culture positive urinary tract infection at baseline assessment, or those with a urine dip positive for leukocytes and nitrates on straight catheterized sample.
* Patients who have received antibiotics within the past two weeks
* Patients with stage 3 or 4 pelvic organ prolapse based on the pelvic organ prolapse quantitation system (POP-q)
* Patients unwilling to use vaginal estrogen preparation
* Patients currently on anticholinergic medications or who have received anticholinergic medications within the past three months
* Patients who have previously failed two medications for treatment of OAB or have previously received more advanced treatment for OAB including intra-vesicle botulinum toxin injections, posterior tibial nerve stimulation, or implantation of a sacral neuromodulator
* Patients wishing to start anticholinergic medication at the initial encounter
* Undiagnosed abnormal genital bleeding
* Active deep vein thrombosis (DVT), pulmonary embolism (PE), or a history of these conditions
* Active arterial thromboembolic disease (for example, stroke and MI), or a history of these conditions
* Known liver dysfunction or disease
* Known protein C, protein S, or antithrombin deficiency or other known thrombophilic disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Wolfe, PhD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearce MM, Hilt EE, Rosenfeld AB, Zilliox MJ, Thomas-White K, Fok C, Kliethermes S, Schreckenberger PC, Brubaker L, Gai X, Wolfe AJ. The female urinary microbiome: a comparison of women with and without urgency urinary incontinence. mBio. 2014 Jul 8;5(4):e01283-14. doi: 10.1128/mBio.01283-14. PMID 25006228
- [Background] Hilt EE, McKinley K, Pearce MM, Rosenfeld AB, Zilliox MJ, Mueller ER, Brubaker L, Gai X, Wolfe AJ, Schreckenberger PC. Urine is not sterile: use of enhanced urine culture techniques to detect resident bacterial flora in the adult female bladder. J Clin Microbiol. 2014 Mar;52(3):871-6. doi: 10.1128/JCM.02876-13. Epub 2013 Dec 26. PMID 24371246
- [Background] Wolfe AJ, Toh E, Shibata N, Rong R, Kenton K, Fitzgerald M, Mueller ER, Schreckenberger P, Dong Q, Nelson DE, Brubaker L. Evidence of uncultivated bacteria in the adult female bladder. J Clin Microbiol. 2012 Apr;50(4):1376-83. doi: 10.1128/JCM.05852-11. Epub 2012 Jan 25. PMID 22278835
- [Background] Khasriya R, Sathiananthamoorthy S, Ismail S, Kelsey M, Wilson M, Rohn JL, Malone-Lee J. Spectrum of bacterial colonization associated with urothelial cells from patients with chronic lower urinary tract symptoms. J Clin Microbiol. 2013 Jul;51(7):2054-62. doi: 10.1128/JCM.03314-12. Epub 2013 Apr 17. PMID 23596238
- [Background] Fouts DE, Pieper R, Szpakowski S, Pohl H, Knoblach S, Suh MJ, Huang ST, Ljungberg I, Sprague BM, Lucas SK, Torralba M, Nelson KE, Groah SL. Integrated next-generation sequencing of 16S rDNA and metaproteomics differentiate the healthy urine microbiome from asymptomatic bacteriuria in neuropathic bladder associated with spinal cord injury. J Transl Med. 2012 Aug 28;10:174. doi: 10.1186/1479-5876-10-174. PMID 22929533
- [Background] Fok CS, McKinley K, Mueller ER, Kenton K, Schreckenberger P, Wolfe A, Brubaker L. Day of surgery urine cultures identify urogynecologic patients at increased risk for postoperative urinary tract infection. J Urol. 2013 May;189(5):1721-4. doi: 10.1016/j.juro.2012.11.167. Epub 2012 Dec 3. PMID 23219547
- [Background] Nelken RS, Ozel BZ, Leegant AR, Felix JC, Mishell DR Jr. Randomized trial of estradiol vaginal ring versus oral oxybutynin for the treatment of overactive bladder. Menopause. 2011 Sep;18(9):962-6. doi: 10.1097/gme.0b013e3182104977. PMID 21532512
- [Background] Tseng LH, Wang AC, Chang YL, Soong YK, Lloyd LK, Ko YJ. Randomized comparison of tolterodine with vaginal estrogen cream versus tolterodine alone for the treatment of postmenopausal women with overactive bladder syndrome. Neurourol Urodyn. 2009;28(1):47-51. doi: 10.1002/nau.20583. PMID 19089890
- [Background] Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, Goldman HB, Huser M, Milani AL, Moran PA, Schaer GN, Withagen MI. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic organ prolapse (POP). Int Urogynecol J. 2016 Apr;27(4):655-84. doi: 10.1007/s00192-016-3003-y. PMID 26984443
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Cardozo LD, Wise BG, Benness CJ. Vaginal oestradiol for the treatment of lower urinary tract symptoms in postmenopausal women--a double-blind placebo-controlled study. J Obstet Gynaecol. 2001 Jul;21(4):383-5. doi: 10.1080/01443610120059941. PMID 12521832
- [Background] Eriksen PS, Rasmussen H. Low-dose 17 beta-estradiol vaginal tablets in the treatment of atrophic vaginitis: a double-blind placebo controlled study. Eur J Obstet Gynecol Reprod Biol. 1992 Apr 21;44(2):137-44. doi: 10.1016/0028-2243(92)90059-8. PMID 1587379
- [Background] Brading AF. A myogenic basis for the overactive bladder. Urology. 1997 Dec;50(6A Suppl):57-67; discussion 68-73. doi: 10.1016/s0090-4295(97)00591-8. PMID 9426752
- [Background] Griebling TL, Liao Z, Smith PG. Systemic and topical hormone therapies reduce vaginal innervation density in postmenopausal women. Menopause. 2012 Jun;19(6):630-5. doi: 10.1097/gme.0b013e31823b8983. PMID 22205148
- [Background] Brotman RM, Shardell MD, Gajer P, Fadrosh D, Chang K, Silver MI, Viscidi RP, Burke AE, Ravel J, Gravitt PE. Association between the vaginal microbiota, menopause status, and signs of vulvovaginal atrophy. Menopause. 2014 May;21(5):450-8. doi: 10.1097/GME.0b013e3182a4690b. PMID 24080849
- [Background] Raz R. Urinary tract infection in postmenopausal women. Korean J Urol. 2011 Dec;52(12):801-8. doi: 10.4111/kju.2011.52.12.801. Epub 2011 Dec 20. PMID 22216390
- [Background] Coyne KS, Thompson CL, Lai JS, Sexton CC. An overactive bladder symptom and health-related quality of life short-form: validation of the OAB-q SF. Neurourol Urodyn. 2015 Mar;34(3):255-63. doi: 10.1002/nau.22559. Epub 2014 Jan 13. PMID 25783168
- [Background] Rahn DD, Ward RM, Sanses TV, Carberry C, Mamik MM, Meriwether KV, Olivera CK, Abed H, Balk EM, Murphy M; Society of Gynecologic Surgeons Systematic Review Group. Vaginal estrogen use in postmenopausal women with pelvic floor disorders: systematic review and practice guidelines. Int Urogynecol J. 2015 Jan;26(1):3-13. doi: 10.1007/s00192-014-2554-z. Epub 2014 Nov 13. PMID 25392183
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435
- [Derived] Thomas-White K, Taege S, Limeira R, Brincat C, Joyce C, Hilt EE, Mac-Daniel L, Radek KA, Brubaker L, Mueller ER, Wolfe AJ. Vaginal estrogen therapy is associated with increased Lactobacillus in the urine of postmenopausal women with overactive bladder symptoms. Am J Obstet Gynecol. 2020 Nov;223(5):727.e1-727.e11. doi: 10.1016/j.ajog.2020.08.006. Epub 2020 Aug 11. PMID 32791124

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Estrogen Arm
Started | 35
Completed | 24
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Estrogen Arm
Number analyzed (Participants) | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [62 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23
  African American | 8
  Asian | 1
  Hispanic | 2
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 35
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.5 [26.0 to 35.9]
Number of vaginal deliveries [Median (Inter-Quartile Range); unit: deliveries] | 3 [2 to 3]
Prior hysterectomy [Count of Participants; unit: Participants]
  Prior hysterectomy | 16
  No prior hysterectomy | 19
Stage of prolapse [Count of Participants; unit: Participants] — Stage was determined using the Pelvic Organ Prolapse Quantification (POP-Q), where higher stage indicates greater degree of prolapse. Those with no prolapse are stage 0. For stage 1, the most distal portion of the prolapse is more than 1 cm above the level of the hymen. For stage 2, the most distal portion of the prolapse is situated between 1 cm above the hymen and 1 cm below the hymen.
  Participants
    0 | 9
    1 | 11
    2 | 15
Ovaries removed [Count of Participants; unit: Participants]
  Ovaries removed | 7
  Ovaries not removed | 26
  Unknown | 2
Previous incontinence surgery [Count of Participants; unit: Participants]
  Previous incontinence surgery | 2
  No previous incontinence surgery | 33
Postvoid residual [Median (Inter-Quartile Range); unit: mL] | 40 [25 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Change in the Relative Abundance of Lactobacillus
Description: The relative abundance of Lactobacillus to total microbes per sample was measured before and after treatment. The within-participant change in relative abundance of Lactobacillus was calculated subtracting pre-treatment from post-treatment.
Time Frame: 0, 12 weeks
Population: Participants with catheterized urine samples taken pre-treatment and post-treatment
Measure: Mean (Standard Deviation); unit: proportion of total microbes
Arm/Group | Estrogen Arm
Number analyzed (Participants) | 18
proportion of total microbes | 0.275 (0.345)

2. Secondary Outcome: Change in OAB Symptoms
Description: OAB symptoms are measured using the Overactive Bladder Questionnaire (OAB-q). The OAB-q symptom score ranges from 0-100 with higher scores indicating greater symptom severity. A change score is calculated as the post-treatment score minus the pre-treatment score.
Time Frame: 0, 12 weeks
Population: All participants who completed the OAB symptoms questionnaire at baseline and after treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Estrogen Arm
Number analyzed (Participants) | 24
units on a scale | -21 [-39 to -8]

3. Secondary Outcome: OAB Symptoms Associated With Relative Abundance of Lactobacillus
Description: The investigators will determine whether change in OAB symptoms using the OAB-q before and after treatment is associated with the change in participants' relative abundance of Lactobacillus before and after treatment. The OAB-q symptom score ranges from 0-100 with higher scores indicating greater symptom severity.
Time Frame: 0, 12 weeks
Population: All participants who completed the OAB symptoms questionnaire and have catheterized urine samples at baseline and after treatment
Measure: Number; unit: Spearman's rho
Arm/Group | Estrogen Arm
Number analyzed (Participants) | 18
Spearman's rho | -0.32

4. Secondary Outcome: Change in Urothelial Antimicrobial Peptide (AMP) Levels
Description: The investigators will compare participants' AMP activity levels before and after treatment. AMP activity level is measured as the diffusion of AMPs in bacterial agar from the center of the well to which the patient's purified biological sample is applied. The diffusion of AMPs in the agar results in the killing of bacteria and a clearing around the well. This clearing of bacterial growth is measured in square millimeters and then normalized to the total peptide concentration. Change is calculated as the post-treatment AMP activity level minus the pre-treatment AMP activity level.
Time Frame: 0, 12 weeks
Population: Assays were performed on a subset of participants due to resource constraints.
Measure: Median (Full Range); unit: normalized bacterial growth inhibition
Arm/Group | Estrogen Arm
Number analyzed (Participants) | 2
normalized bacterial growth inhibition | 0.14 [0.07 to 0.22]

5. Secondary Outcome: Change in OAB Symptoms Associated With Change in AMP Levels
Description: The investigators will determine whether any change in OAB symptoms using the OAB-q before and after treatment is associated with the change in participants' AMP levels before and after treatment.
Time Frame: 0, 12 weeks
Population: Assays were performed on a subset of participants due to resource constraints.
Measure: Number; unit: Spearman's rho
Arm/Group | Estrogen Arm
Number analyzed (Participants) | 2
Spearman's rho | -1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Estrogen Arm
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT02835846/Prot_SAP_000.pdf